# OFFICIAL TITLE OF STUDY:

Statewide Implementation of CAPABLE-Community Aging in Place, Advancing Better Living for Elders in the Michigan Medicaid Home and Community Based Waiver Program

> NCT NUMBER: NCT03634033 Registered August 16, 2018

DOCUMENT DATE: FEBRUARY 4, 2019



## **Research Study**

**Title:** Statewide Implementation of CAPABLE (Community Aging-in-Place, Advancing Better Living for Elders) in the Michigan Medicaid Home and Community Based Waiver Program (NIA1R15AG058193-01A1S1; NCT03634033)

Researcher: Sandra L. Spoelstra

You are being asked to participate in a research study. The box below highlights key information about this research study for you to consider when making a decision whether or not to participate. Carefully consider this information and the additional information on this form. Please ask questions about any of the information you do not understand before you decide whether to participate.

## **Key Information for You to Consider**

**Voluntary Consent.** You are being asked to volunteer for this research study. It is up to you whether you choose to participate or not. If you choose NOT to participate, there are instructions below on how to opt out of the research. Opting out will <u>NOT</u> affect employment status.

**Purpose**. This is a collaborative research effort between the Grand Valley State University College of Nursing, the State of Michigan Department of Health and Human Services, and the National Institutes of Aging to find out if different supervisory procedures add to how well CAPABLE works to help participants stay at home and in the community.

**Duration**. It is expected that your participation will last one year.

**Procedures and Activities.** You will complete a survey asking you about your characteristics and your waiver site leadership and readiness to implement CAPABLE. You will complete training on CAPABLE and a survey asking you about your attitude, self-efficacy, and knowledge of and satisfaction with training. Throughout the study, you will conduct CAPABLE with your participants in addition to usual waiver care services. At the end, you will complete a survey asking about your attitude and self-efficacy.

**Risks**. It is not expected that you will be placed at any physical, financial, or legal risk or harm to your employment status as a result of taking part in this study.

**Benefits**. There are no direct benefits to you, but we believe the knowledge gained from this study will increase clinician knowledge regarding CAPABLE and assist waiver sites to care for their participants. **Alternatives**. Participation is voluntary and if you choose to opt out, your employment will not be affected.

# How will this study help me?

Information from this study may help researchers understand how to help participants stay in their home longer, increase clinician knowledge regarding CAPABLE, and assist waiver sites to care for participants, who may experience improved function, pain, falls, depression, and reduced hospitalizations and emergency room visits.

# Who can participate?

We are inviting all Supports Coordinators, who are 21 years of age or older, and have chosen NOT to opt out of this study.

## What will you receive?

If you agree to take part of the study:

■ You will complete an online survey (10-20 minutes) asking you about your characteristics and your waiver site leadership and readiness to implement CAPABLE.

- You will complete an online training (4-6 hours) on CAPABLE and survey questions (5-10 minutes) asking you about your characteristics, attitude, self-efficacy, and knowledge of and satisfaction with training.
- Throughout the study's duration, you will conduct CAPABLE with your participants in addition to "usual" waiver care services.
- At the end of the study, you will complete an online survey (20-30 minutes) asking about your attitude and self-efficacy.

#### What information will be used for research?

We will be collecting your data within an online survey platform (Qualtrics). This will include information about your discipline, how long you worked in the waiver, and your self-efficacy, belief about evidence, and readiness for change. We will have your name in order to follow your progress, but this information is known ONLY to the researcher and will be stored on a secure server. To prevent your identity to be connected with your data, we will remove specified individual identifiers (e.g. names, phone numbers, etc.) from the data. NO private information will be shared with anyone other than the researcher, and your results will be pooled among the other participants.

#### Are there risks?

It is not expected that you will be placed at any physical, financial, or legal risk or harm to your employment status as a result of taking part in this study. A Certificate of Confidentiality has been obtained from the Department of Health and Human Services for this study. To help protect your privacy, this certificate prevents researchers from being required (subpoenaed) to disclose identifying sensitive information collected for this study for use in court in most cases."

• If you have questions about the research study call: Sandra Spoelstra, Grand Valley State University, at 616-331-5905

#### What do I have to do?

If you are willing to let us use your information to better understand how well the program is working, you do not have to do anything, as you will be included in the study.

If you wish to NOT have your information used, you can opt out of the study. Your decision to participate or not will not affect your current or future employment.

To opt out and NOT have your information used, please contact the researcher via phone:

Sandra Spoelstra at Grand Valley State University at 616-331-5905.

## What if I change my mind during the study?

You are free to change your mind at any time and you may withdraw from the study if you like by calling Sandra Spoelstra at 616-331-5905. We will remove your data from our study.

If you have any questions about your rights as a research participant, please contact the Office of Research Compliance & Integrity at Grand Valley State University, 1 Campus Dr., Allendale, MI Phone 616-331-3197. E-mail: rci@gvsu.edu

This study was approved by the Grand Valley State University Human Research Review Committee (Protocol 19-061-H) on XX/XX/XXXX.